CLINICAL TRIAL: NCT03644498
Title: Risk of Muscle Damage in Cancer Patients Exposed to the Influenza Vaccine While Receiving Checkpoint Inhibitor Therapies: A Nested Case Control Study Using Claims Data
Brief Title: Study to Determine if the Flu Vaccine Increases the Risk of Muscle Damage in Participants Taking Drugs That Block Certain Proteins Made by Some Types of Immune System Cells
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-99J
Record Dates: First submitted 2018-08-22; First posted 2018-08-23 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Cancer
Keywords: influenza; myositis; myocarditis; rhabdomyolysis; checkpoint inhibitors
MeSH Terms: conditions — Neoplasms; Influenza, Human; Myositis; Myocarditis; Rhabdomyolysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults treated with a CPI therapy for cancer
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
A retrospective, observational study conducted on cancer patients receiving a drug that blocks certain proteins made by some types of immune system cells

ELIGIBILITY:
Inclusion Criteria:

* Treatment with a checkpoint inhibitor (CPI)
* Age greater than or equal to 18 years on date of first claim for a CPI
* ICD-9 or ICD-10 code for a malignancy within 180 days prior to the first claim for any CPI, and
* Greater than or equal to 180 days of continuous pharmaceutical and medical benefit enrollment in the database prior to the first claim for any CPI

Exclusion Criteria:

* Less than 18 years of age

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants in this study will be enrolled in the PharMetrics or MarketScan database and will have exposure to at least one checkpoint inhibitor
Sampling Method: Probability Sample
Enrollment: 1056 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2018-10-17 (Actual)

PRIMARY OUTCOMES:
Incidence of myocarditis | Approximately 7 years
Incidence of myositis | Approximately 7 years
Incidence of rhabdomyolysis | Approximately 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Princeton, New Jersey, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html